CLINICAL TRIAL: NCT06481956
Title: Phase II Clinical Study of Trastuzumab Emtansine (T-DM1) Combined With Cyclin-dependent Kinase 4/6 (CDK4/6) Inhibitor Ribociclib in the Treatment of Human Epidermal Growth Factor Receptor-2 (HER2)-Positive Advanced Breast Cancer
Brief Title: T-DM1 Combined With CDK4/6 Inhibitor Ribociclib
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Zheng Yabing (Other)
Responsible Party: Sponsor-Investigator, Zheng Yabing, Deputy director, Zhejiang Cancer Hospital
Organization: Zhejiang Cancer Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: [2023]-06-10
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: HER2-positive Advanced Breast Cancer
Keywords: HER2-positive; Advanced breast cancer; Trastuzumab Emtansine; Ribociclib
MeSH Terms: interventions — ribociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- T-DM1 combined with Ribociclib (Experimental): Enrolled patients will receive (repeat every 21 days) :
  ● T-DM1 3.6 mg/kg d1;● Ribociclib 400 mg qd, d8-d21;
  * ER-positive patients will receive endocrine therapy at the same time: aromatase inhibitors or fulvestrant , and ovarian suppression or ovariectomy in premenopausal women.
  Interventions: Drug: Ribociclib Oral Tablet

INTERVENTIONS:
Drug: Ribociclib Oral Tablet — Patients with advanced breast cancer with at least one evaluable lesion and histologically proven invasive breast cancer were eligible for inclusion. Histopathologically positive for HER2 (IHC 3+, or IHC 2+ with fluorescence in situ hybridization (FISH) positive, either primary or metastatic. Patients with advanced breast cancer must have previously received first-line therapy or initial rescue therapy and have been treated with trastuzumab against HER2.

SUMMARY:
To explore the efficacy and safety of T-DM1 combined with CDK4/6 inhibitor Ribociclib in the treatment of HER2-positive advanced breast cancer.

DETAILED DESCRIPTION:
This is a multicenter, single-arm,Phase II clinical trial to explore the efficacy and safety of Trastuzumab Emtansine (T-DM1) combined with CDK4/6 inhibitor Ribociclib in the treatment of unresectable locally advanced or metastatic HER2-positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 at the time of signing the informed consent.
* Patient's ability to follow the study protocol as determined by the investigator.
* A representative tumor tissue sample is required to confirm a HER2-positive diagnosis.

HER2 expression status and ER expression status of invasive cancer lesions were determined based on previous pathological sections or current pre-treatment biopsy materials, and the HER2 IHC assay was locally confirmed to be consistent with 3+, or IHC assay with 2+, and further FISH detection was positive before study enrollment.

* At least one evaluable lesion was detected by CT or MRI (see protocol for additional details).
* For metastatic or recurrent breast cancer, there is currently no opportunity for surgical radical resection.
* Metastatic or recurrent breast cancer that has received at least first-line rescue therapy in the past must have been treated with trastuzumab and taxanes.
* The Physical status (ECOG) score of the Eastern Tumor Collaboration group was 0 or 1.
* Sufficient haematology and organ function to meet the definition of laboratory test results, which must be provided within 14 days before the start of study therapy.
* Fertile women should remain abstinent (no heterosexual intercourse) or use contraceptive methods.

Exclusion Criteria:

* Past treatment with other antibody-drug conjugate (ADC) drugs or anti-tumor therapy with CDK4/6 inhibitors.
* Past treatment with other anti-HER2 drugs other than trastuzumab, pertuzumab and tyrosine kinase inhibitors (TKI).
* Advanced breast cancer with central nervous system metastasis.
* Patients who have developed other malignancies in the 5 years prior to screening, except adequately treated cervical cancer in situ, non-melanoma skin cancer, localized prostate cancer, ductal carcinoma in situ, or stage I uterine cancer.
* Severe dysfunction of vital organs prior to enrollment (see protocol details).
* Received an investigational drug within 28 days prior to initiation of study therapy.
* Known hypersensitivity or hypersensitivity to CDK4/6 inhibitors.
* The results of the serum pregnancy test were positive.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2027-01-10 (Estimated); Study Completion 2027-10-10 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to 54 months
  ORR is defined as the percentage of patients who achieved a best overall response of Complete Response (CR) or Partial Response (PR), per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1) for target lesions as assessed by the Investigator: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | up to 54 months
  From date of first dose until the date of first documented progression or date of death from any cause, whichever came first.
2-year Overall Survival (OS) | up to 54 months
  the overall survival rate in all patients from the date of first dose to the end of follow-up at 2 years.
Objective Response Rate of Subgroup Population (ORR) | up to 54 months
  Objective Response Rate of subgroup population (ER>=10% vs ER<10%)
Adverse Event (AE) | up to 54 months
  Evaluation performed using the National Cancer Institute (NCI)- Standard for Common Terminology for Adverse Events (CTCAE)v.5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Yabing Zheng, MD, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China